CLINICAL TRIAL: NCT02025517
Title: Immediate Effects of Treadmill Gait Training Combined With Cognitive Tasks in Individuals With Parkinson's Disease: Randomized Controlled Trial
Brief Title: Gait Training With Cognitive Tasks in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Ana Raquel Rodrigues Lindquist, Ana Raquel Rodrigues Lindquist, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEP-UFRN 03063812.0.0000.5537
Record Dates: First submitted 2013-12-13; First posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2012-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; rehabilitation; kinematics; cognition
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Without Cognitive Tasks (No Intervention): Gait training on treadmill during 20 minutes.
- Cognitive Tasks (Experimental): Treadmill training plus cognitive verbal fluency, memory and spatial planning tasks, during 20 minutes.
  Interventions: Other: Cognitive Tasks.

INTERVENTIONS:
Other: Cognitive Tasks. — The Experimental Group underwent treadmill gait training simultaneously to a protocol of cognitive tasks created specifically for this study, based on cognitive activities proposed in previous studies. The training sessions lasted 20 minutes. The first three minutes allowed subjects to familiarize themselves with the treadmill. From the 4th minute onward, the volunteer walked for 1 minute while performing cognitive tasks, and in the following minute, only walked. Thus, the 17 remaining minutes on the treadmill alternated between one minute of treadmill training combined with a cognitive task and the following minute only treadmill training. Treadmill gait speed was that reported by the patient as the fastest possible speed while maintaining a suitable comfort level.
  Arms: Cognitive Tasks

SUMMARY:
Treadmill gait training combined with cognitive tasks in Parkinson's disease.

DETAILED DESCRIPTION:
This is a trial involving subjects diagnosed with Parkinson's disease, in accordance with guidelines established by the London Brain Bank.

Individuals often must execute more than one task simultaneously during everyday life. When different activities that require attention are performed at the same time, a situation called Dual Task occurs.

Under normal conditions, motor cortex areas (primary motor cortex, pre-motor cortex and supplementary motor area) are responsible for selecting the range of movements in a given action sequence, in accordance with the demands of the task and environmental restrictions, and after the onset of movements brought about by the motor cortex, the basal nuclei continue execution, leaving the motor cortex free for other tasks that require attention. However, in Parkinson's disease, automaticity promoted by basal nuclei is compromised and constant conscious control becomes necessary during gait. Thus, when an activity concurrent with this function is performed, the frontal regions become dedicated to the secondary task and gait is predominantly controlled by defective basal nuclei, which generates negative Dual Task interference on gait.

Given the poor gait quality assessed in DT situations, individuals with PD have been instructed to avoid these circumstances. By contrast, recent evidence has demonstrated that gait training in conjunction with to secondary activities is capable of improving variables related to DT gait performance in PD.

Considering that treadmill gait training provides greater regularity and automaticity, allowing subjects to divert their attention to cognitive functions, this study hypothesizes that DT treadmill gait training combined with cognitive tasks will promote better gait performance in individuals with PD.

Patients were invited to participate in the study from phone calls. They were recruited from the service list in Neurology at Hospital Onofre Lopes, in Natal -Brazil. Randomization of individuals with respect to participation in the groups was done via the randomization.com website, by a person unfamiliar with the training procedures (rater 1), who assigned a color (yellow or green) to each group. Opaque envelopes were numbered and separated, and inside each envelope was a piece of paper containing the word "yellow" or "green". As a new patient arrived for training, rater 2 opened an envelope and was only aware of the color code of that particular patient. Rater 3, the lead researcher, conducted the assessment and re-assessment procedures. The color codes were maintained in secrecy by raters 1 and 2 throughout the entire study.

Cognitive function was assessed using the Montreal Cognitive Assessment Scale (MoCA). Its score ranges between 0 and 30, covering aspects related to visuospatial and executive functions, naming, memory, attention, language, abstraction, delayed recall, as well as temporal and spatial orientation. Higher scores correspond to greater cognitive function.

Disease severity was classified according to guidelines proposed by the Modified Hoehn and Yahr Scale, composed of seven stages, allowing categorization of both sides of the body as to balance and physical independence. Its scores range from 0 (no signs of the disease) to 5 points (confined to bed or wheelchair).

Assessment of degree of motor and functional impairment was obtained using the Unified Parkinson's Disease Rating Scale (UPDRS). This study used only items 2 and 3 of the scale, related to ADLs and motor exploration, whose scores correspond to 52 and 56, respectively.

Kinematic assessment of overground gait was performed by the Qualisys Motion Capture Systems (Qualisys Medical AB, 411 13 Gothenburg, Sweden), which records the spatiotemporal variables of gait, as well as angular variations of hip, knee and ankle joints. This system is composed of eight cameras that emit and capture infrared light. The light is reflected by spherical passive markers positioned on bony prominences and standard body segments, in order to capture lower limb data. The cameras are connected to a computer, where the images collected are stored. Data captured in two-dimensional imaging are processed by Qualisys Track Manager 2.6 acquisition software, which recognizes marker positioning and, based on the combination of images from at least two cameras connected in series, enables the generation of three-dimensional coordinates of movement. To that end, data are transported by 3D visual software (C-Motion, Rockville, MD, USA), version Basic/RT 3.99.25.8), which allows the reconstruction and three-dimensional analysis of the body segments marked, thereby recording the movements executed during gait.

For kinematic assessment, we used 15 and 19 mm-diameter markers positioned bilaterally on the following structures: iliac crest, greater trochanter, medial and lateral epicondyle of the femur, medial and lateral malleoli, calcaneus, head of the first metatarsal and head of the fifth metatarsal. These markers are denominated anatomical, since their function is to demarcate axial joints, allowing different segments to be delimited.

The marks that guide the trajectory of segments are classified as tracking, and are arranged in fours on the rectangular base (cluster). The markers were placed on the base of the sacrum, on the middle third of the thigh and middle third of the leg. Anatomical markers were fixed with double-faced adhesive tape and reinforced with surgical tape, while tracking markers were coupled to the body segments with elastic bands and Velcro. Markers were colored by the same rater on all the volunteers, in order to preserve the reliability of the marking.

For gait training, we used an electric Gait Trainer 2 treadmill (Biodex Medical System, NY, USA), with a walking area measuring 160 x 51 centimeters (cm), and equipped with a bar for upper extremity support, heart monitoring by bioimpedance sensors located on the bar and a Polar Telemetry system (POLAR, USA). Coupled to the treadmill is an Unweighing System (Biodex Medical System, NY, USA), composed of a vertical standing frame that carries the weight supported by means of a harness. However, the patients did not use the weight support system in this study and the harness was used only as a safety precaution during the training sessions.

The study procedures were performed over two days, the first for assessment and the second for the intervention with immediate reassessment. On the first day, the Montreal Cognitive Assessment (MoCA), Unified Parkinson's Disease Rating Scale and Modified Hoehn and Yahr Scale were applied. Next, weight and height were recorded. Finally, kinematic assessment of overground DT gait was carried out. On the second day, the subjects were submitted to treadmill training and kinematic reassessment of overground DT gait. Assessment occurred one day after training.

At the onset of kinematic assessment, after marker placement and equipment calibration, static collection was performed to inform the system regarding body segment positioning and enable subsequent construction of the biomechanical model. The individual remained in the orthostatic position, with arms crossed over their chest, feet apart and pointing towards one of the cameras. Subjects were filmed for 3 seconds in this position. Next, the anatomical markers were removed in order to perform dynamic captures. Only tracking markers of thigh and leg segments remained in place, as well as those on the head of the fifth metatarsal, lateral malleolus and calcaneus, which correspond to the foot segment.

At each dynamic capture, the individuals were instructed to cover a distance of 8 meters, walking at maximum speed, while performing a cognitive task. During each 8-meter lap a letter was randomly drawn and the individual was asked to say as many words as possible starting with that letter. When the patients unable to recall words, the subjects were also instructed not to stop, but rather to continue walking and trying to remember. Ten dynamic collections were conducted.

On the next day, the Experimental Group (n=11) underwent treadmill gait training simultaneously to a protocol of cognitive tasks involving a number of attention and executive functions, such as verbal fluency, working memory and spatial planning. The protocol was created specifically for this study, based on cognitive activities proposed in previous studies. The training sessions lasted 20 minutes. The first three minutes allowed subjects to familiarize themselves with the treadmill. From the 4th minute onward, the volunteer walked for 1 minute while performing cognitive tasks, and in the following minute, only walked. Thus, the 17 remaining minutes on the treadmill alternated between one minute of treadmill training combined with a cognitive task and the following minute only treadmill training. The Control Group (n=11) underwent only treadmill training. Training lasted 20 minutes for both groups. Treadmill gait speed for both groups was that reported by the patient as the fastest possible speed while maintaining a suitable comfort level. Vital signs (heart rate and blood pressure) were monitored before, during and after the session.

Immediately after treadmill training, DT overground gait was reassessed, using ten dynamics captures, the same procedures used on the first day.

Kinematic data processing was conducted with Qualisys Track Manager 2.6 software (QTM), where markers were named and their trajectories defined. Next, the data obtained in QTM were exported to the Visual 3D program, where three-dimensional reconstruction of the biochemical model was carried out.

Statistical analysis was conducted using the Statistical Package for the Social Sciences (SPSS), version 19.0. Before the analysis of each group, data distribution normality was verified by applying descriptive statistics procedures and the Kolmogorov-Smirnov (K-S) test.

Measures of central tendency and dispersion were used to illustrate clinical, demographic and anthropometric data. For data with normal distribution, the paired t-test was used to compare intragroup spatiotemporal and angular variables, while the student's t-test for independent samples was applied to compare intergroup variables. The Mann-Whitney test was used for data with non-normal distribution. A significance level of 5% was set for all these tests.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD by a neurologist and confirmed by complementary examinations;
* Degree of disease progression equivalent to stages 2 to 3 of the Modified Hoehn and Yahr Scale;
* Regular use of antiparkinson medication, exhibiting stable response; able to walk independently without ortheses or other assistive devices;
* Absence of brain stimulation surgery; absence of cardiovascular, respiratory and musculoskeletal diseases that could compromise performance during assessment and training;
* Absence of other neurological disorders;
* Absence of non-corrected visual or auditory disturbances;
* Be able to understand verbal instructions; being literate;
* Give their written informed consent.

Exclusion Criteria:

* Blood pressure above 140X90 mmHg before the intervention (values referring to the first stage of hypertension);
* Heart rate above the submaximal value, calculated by the formula 0.75 x (220-age), during the intervention;
* Feeling nauseous or experiencing persistent acute pain during the exercises; - Voluntarily abandoning the study.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Changes in kinematic gait parameters after treadmill training | Immediately after gait training on treadmill.
  The treadmill training was realized for 20 minutes. Immediately after treadmill training, kinematic gait data were captured by Qualisys Track Manager software and exported to Visual 3D, to reconstruct the segments and create a biomechanical model. It was carried out in two stages: static and dynamic collection. The primary outcome measure was the kinematic variables at the phase post training on treadmill. The kinematic variables include: speed (m/s), cadence (steps/min), stride length (m), step length (m) and angular displacement (º).

CONTACTS AND LOCATIONS:
Overall Officials: Angelica VC Sousa, Master, Principal Investigator — Universidade Federal do Rio Grande do Norte
Locations (1):
- Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil